CLINICAL TRIAL: NCT06429956
Title: Combining Treatment Components in Transdiagnostic Therapy for Anxiety and Depression: A Randomized Controlled Trial
Brief Title: Combining Treatment Components in Transdiagnostic Therapy for Anxiety and Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Combinatory effects in CBT 24
Record Dates: First submitted 2024-05-13; First posted 2024-05-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either 1) the mindful emotion awareness module followed by the cognitive flexibility module or 2) the cognitive flexibility module followed by the mindful emotion awareness module. All participants will undergo a three-week waiting period before starting treatment.
Who Masked: Participant
Masking Description: It will not be known to participants that we are testing combinatory and sequencing effects and that participants are randomly allocated to receive the treatment modules in a specific order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Order 1 (mindful emotion awareness + cognitive flexibility) (Experimental): Participants will receive 6 therapy sessions starting with 3 sessions of mindful emotion awareness followed by 3 sessions of cognitive flexibility. Each session will have a duration of approximately 1 hour. Treatment will follow the UP manual by Barlow et al. (2018).
  Interventions: Behavioral: Mindful emotion awareness; Behavioral: Cognitive flexibility
- Order 2 (cognitive flexibility + mindful emotion awareness) (Experimental): Participants will receive 6 therapy sessions starting with 3 sessions of cognitive flexibility followed by 3 sessions of mindful emotion awareness. Each session will have a duration of approximately 1 hour. Treatment will follow the UP manual by Barlow et al. (2018).
  Interventions: Behavioral: Mindful emotion awareness; Behavioral: Cognitive flexibility

INTERVENTIONS:
Behavioral: Mindful emotion awareness — The mindful emotion awareness module will follow the manual by Barlow et al. (2018). In session 1, the participant will receive psychoeducation about the purpose of mindful emotion awareness (i.e., to cultivate present-focused, non-judgmental attention to one's emotional experiences) and will complete an in-session guided meditation exercise which they will be asked to practice daily using an audio file. In session 2 and 3, two additional exercises are introduced. With "mindful mood induction", the participant is instructed to induce emotions and then practice mindful emotion awareness in this context. With "anchoring in the present", the participant is taught four steps to help them use mindful emotion awareness to pull themself back to the present whenever they feel an emotional response start to build in their everyday life. For homework, the participant will practice mindful emotion using these exercises and the audio file.
Behavioral: Cognitive flexibility — The cognitive flexibility module will follow the manual by Barlow et al. (2018) which is based on the principles by Beck (1976). In session 1, the participant will be psychoeducated about the purpose of cognitive flexibility (i.e., to encourage flexible thinking through reappraisal of one's automatic thinking), and how their thoughts influence their emotional reactions. For homework, the participant will be asked to monitor their automatic thoughts. In session 2, the participant will be introduced to the technique of cognitive flexibility (i.e., generating other possible interpretations), and this technique will be practiced throughout session 2 and 3. For homework, the participant will continue to monitor their automatic thoughts and generate and record other possible interpretations.

SUMMARY:
The present study is a randomized controlled trial that will evaluate the effect of combining two treatment components (i.e., cognitive restructuring and detached mindfulness) drawn from cognitive behavioral therapies (CBTs) that are often combined in clinical practice. However, knowledge about the effect of combining these treatment components is lacking. Therefore, this study aims to explore single, combined, and sequencing effects of these two treatment components in patients with depression and/or anxiety disorders. Furthermore, the study aims to explore possible demographic and clinical moderators of the effects to address the question of what works for whom.

DETAILED DESCRIPTION:
A relatively large proportion of psychotherapists endorse practicing eclectic or integrative therapy, drawing from different schools of therapy (Norcross & Alexander, 2019). This tendency towards integrative therapy has been expressed by former president of the Association of Cognitive and Behavioral Therapies, J. B. Persons, who writes: "We [clinicians] rarely proceed through a single protocol from beginning to end. Instead, we use what might be called a mix-and-match strategy, in which we select interventions or modules from one or even two or more protocols that we believe will be helpful to the patient" (Persons, 2005, p. 107). Indeed, there has been a growing research and clinical interest in personalized therapy where treatment components from different therapies are combined with the aim of targeting the symptomatology and theorized maintenance processes of the individual patient (Cohen et al., 2021; DeRubeis et al., 2014; Fisher et al., 2019; Fisher & Boswell, 2016; Hayes et al., 2022; Huibers et al., 2021; Sauer-Zavala et al., 2022). In addition to this, an increasing number of therapies are designed by combining components from different treatment models (e.g., modular and process-based therapies; Barlow et al., 2018; Hofmann & Hayes, 2019; Hofmann et al., 2021). As a result, patients are likely to be the recipients of several different techniques or strategies, based on different theoretical models, emphasizing different change principles. However, the extent to which compatibility exists between different treatment components remains an underexplored scientific question. The present study aims to fill this gap.

Combining cognitive behavioral therapies

Cognitive behavioral therapies (CBTs) are among the most well-researched psychological treatments for anxiety and depressive disorders (Cuijpers, 2017; Cuijpers et al., 2014). While CBT is often viewed as one of the major schools of psychotherapy, specific CBTs differ in their rationale and understanding of the key maintaining processes in psychopathology (Hayes, 2004). A core tenet of traditional CBT, also known as second-wave CBT, is that psychopathology is maintained by maladaptive or irrational thoughts (Beck, 1976). Thus, a commonly used therapeutic component derived from second-wave CBT is cognitive restructuring, where the patient is taught to think more realistically about emotion-evoking situations (Beck et al., 1979; Clark & Beck, 2010). Thus, cognitive restructuring can be said to target the content of thoughts.

In contrast, newer contemporary or so-called third-wave CBTs such as metacognitive therapy (MCT), acceptance and commitment therapy (ACT), and mindfulness-based cognitive therapy (MBCT) target thought processes (Hayes, 2004). A commonly used therapeutic component across third-wave CBTs involves teaching the patient to meet their experiences with mindfulness and acceptance rather than attempting to change their form (termed detached mindfulness in MCT, defusion in ACT, and decentering in MCT; Hayes et al., 2012; Segal et al., 2002; Wells, 2009). Thus, it can be argued that second- and third-wave CBTs reflect very different ways of approaching one's inner life.

Despite the differences between second- and third-wave CBTs, treatment components from each wave are often combined. One example of this is the widely employed Unified Protocol (UP) which is a transdiagnostic modular cognitive-behavioral treatment for emotional disorders (e.g., anxiety and depression) (Barlow et al., 2018). In UP, patients are asked to engage in cognitive restructuring (within the treatment module of cognitive flexibility) in one module and to practice detached mindfulness (within the treatment module of mindful emotion awareness) in another (Barlow et al., 2018). Several studies have documented that UP is an effective treatment for anxiety and depression (Longley & Gleiser, 2023). However, since the treatment modules in UP are rooted in different therapeutic traditions with different rationales, an intriguing question remains whether the treatment modules are in fact compatible. If not, then it is possible that UP is effective not because but rather despite the combination of the treatment modules (O'Toole et al., 2024).

Compatibility of components

Regarding the combination of mindful emotion awareness and cognitive flexibility, it is theoretically plausible that these modules might be incompatible since the technique of noticing and accepting one's thoughts/emotions (in the module mindful emotion awareness) could be argued to be in opposition to the technique of actively changing one's thoughts (in the module cognitive flexibility). This notion is supported by a small study (N=12) by Gkika and Wells (2015) which investigated the effect of cognitive restructuring and detached mindfulness in an anxiety-provoking situation in patients with elevated symptoms of social anxiety. They found that each technique alone reduced symptoms of social anxiety. However, when combined, a sequencing effect emerged where detached mindfulness followed by cognitive restructuring, but not the reverse, led to increased anxiety (Gkika & Wells, 2015). Borlimi et al. (2019) similarly demonstrated a sequencing effect. They asked non-clinical participants (N=35) to recall an unpleasant experience and apply either cognitive restructuring or an acceptance technique. Acceptance reduced sympathetic reactivity (i.e., galvanic skin response) more than cognitive restructuring, and importantly, the effect was significantly larger when acceptance followed cognitive restructuring than vice versa (Borlimi et al., 2019).

The studies by Gkika and Wells (2015) and Borlimi et al. (2019) are both laboratory experimental studies. The question thus remains whether and how their findings can be generalized to a clinical context with longer duration of each treatment component. Only one larger intervention study exploring combinatory and sequencing effects exists. In this study, Brose et al. (2023) investigated the effect of internet-based cognitive restructuring and behavioral activation on symptoms of depression delivered over 6 weeks. Individuals with mild to moderate depressive symptoms (N=2,304) were randomized to one of two treatment arms, one receiving behavioral activation followed by cognitive restructuring, the other vice versa. The groups had similar dropout rates and showed similar improvements over time, indicating no incongruency between those two components. Besides differences in size and setting (experimental vs. actual treatment), the study by Brose et al. (2023) also differs from the other clinical studies by testing a "cognitive" component against a "behavioral" component instead of comparing different "cognitive" components (e.g., cognitive restructuring and detached mindfulness) against each other. In this case, the rationales may be more consistent with each other.

Taken together, the research findings described above, coupled with results from the few other available studies of combinatory effects (Dibbets et al., 2012; Woelk et al., 2022), testify that combining otherwise effective stand-alone treatment components 1) does not necessarily yield an additive effect, 2) may even sometimes detract from a positive outcome, and 3) that the combined effect may depend on the order of the components. Thus, to be able to combine different treatment components for anxiety and depression effectively, there is a need for intervention studies examining single, combined, and sequencing effects for treatment components from different therapies that are often combined. Currently, such research is sparse, thereby motivating the present study. Moreover, understanding for whom these effects are likely to occur is important for the appropriate adaptations of therapeutic interventions to fit the needs of the individual patients (i.e., personalized therapy; Cohen et al., 2021).

Aims and hypotheses

The primary aim of the present study is to explore the effect of combining treatment components drawn from different CBTs. Thus, we will explore single, combined, and sequencing effects of two treatment modules (i.e., mindful emotion awareness and cognitive flexibility). These modules are routinely delivered together in UP for patients with anxiety disorders or MDD. It is hypothesized that both mindful emotion awareness and cognitive flexibility, when delivered individually, will be effective in reducing symptoms of anxiety and depression. The study will take an exploratory stance regarding combined and sequencing effects and will explore if combined effects are best understood as non-additive, additive, synergistic or antagonistic (cf. O'Toole et al., 2024).

A secondary aim of the study is to explore possible demographic and clinical moderators of the effects (e.g., primary diagnosis, baseline cognitive function and symptomatology) to address the question of what works for whom.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. A diagnosis of an anxiety disorder (generalized anxiety disorder, social anxiety disorder, or panic disorder with or without agoraphobia) and/or mild to moderate major depressive disorder (MDD) according to DSM-5 (American Psychiatric Association, 2022).
3. Danish language proficiency.
4. Ability and willingness to give informed consent.
5. No or stable antidepressant/antianxiety medication (i.e., same dosage for ≥ 8 weeks).
6. Access to either a smartphone, tablet, or computer with video camera.

Exclusion Criteria:

1. Severe depression deemed to require more intense psychotherapy or medication.
2. Persistent depressive disorder (i.e., depressive symptoms have persisted for 2 years or more).
3. Non-stabilized medication (see above).
4. Currently receiving other psychotherapy or counseling.
5. Not capable of participating online.
6. Lack of Danish proficiency.
7. A history of bipolar disorder.
8. Current or past psychosis.
9. Substance abuse or dependence judged to require treatment.
10. Suicide risk requiring immediate hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms (PHQ-9) | Development from pre-treatment to post-treatment (6 weeks)
  Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001; Spitzer et al., 1999; Spitzer et al., 2000).
Anxiety symptoms (BAI) | Development from pre-treatment to post-treatment (6 weeks)
  Beck's Anxiety Inventory (BAI; Beck et al., 1988; Beck & Steer, 1991).
Symptoms of generalized anxiety disorder (GAD-7) | Development from pre-treatment to post-treatment (6 weeks)
  The General Anxiety Disorder-7 (GAD-7; Spitzer et al., 2006).
Symptoms of social anxiety disorder (SIAS) | Development from pre-treatment to post-treatment (6 weeks)
  The Social Interaction Anxiety Scale (SIAS; Mattick & Clarke, 1998).
Symptoms of panic disorder (PDSS-SR) | Development from pre-treatment to post-treatment (6 weeks)
  The Panic Disorder Severity Scale - Self-Report Version (PDSS-SR; Houck et al., 2002).

SECONDARY OUTCOMES:
Depressive symptoms (PHQ-9) | Development from pre-treatment through 3-month follow-up
  Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001; Spitzer et al., 1999; Spitzer et al., 2000).
Anxiety symptoms (BAI) | Development from pre-treatment through 3-month follow-up
  Beck's Anxiety Inventory (BAI; Beck et al., 1988; Beck & Steer, 1991).
Symptoms of generalized anxiety disorder (GAD-7) | Development from pre-treatment through 3-month follow-up
  The General Anxiety Disorder-7 (GAD-7; Spitzer et al., 2006).
Symptoms of social anxiety disorder (SIAS) | Development from pre-treatment through 3-month follow-up
  The Social Interaction Anxiety Scale (SIAS; Mattick & Clarke, 1998).
Symptoms of panic disorder (PDSS-SR) | Development from pre-treatment through 3-month follow-up
  The Panic Disorder Severity Scale - Self-Report Version (PDSS-SR; Houck et al., 2002).
Quality of life (WHO-5) | Development from pre-treatment to post-treatment and development from pre-treatment through 3-month follow-up
  The World Health Organization (WHO)-5 questionnaire (Bech, 1999; Topp et al., 2015).
Rumination (RRS brooding subscale) | Development from pre-treatment to post-treatment and development from pre-treatment through 3-month follow-up
  The Ruminative Response Scale (RRS) brooding subscale (Treynor et al., 2003).
Worry (PSWQ) | Development from pre-treatment to post-treatment and development from pre-treatment through 3-month follow-up
  The Penn State Worry Questionnaire (PSWQ; Meyer et al., 1990).
Worry (AWS) | Session by session development during the 6 weeks of active treatment
  For in-session questionnaires, the Ambulatory Worry Scale (AWS; Kramer et al., 2021) will be used because it has been specially developed to evaluate state variations in worry.
Decentering (EQ decentering subscale) | Development from pre-treatment to post-treatment and development from pre-treatment through 3-month follow-up
  The Experiences Questionnaire (EQ) decentering subscale (Fresco et al., 2007).
Reappraisal (ERQ) | Development from pre-treatment to post-treatment and development from pre-treatment through 3-month follow-up
  Emotion Regulation Questionnaire (ERQ) reappraisal subscale (Gross & John, 2003).
Mindfulness (FFMQ-15) | Development from pre-treatment to post-treatment and development from pre-treatment through 3-month follow-up
  Five Facet Mindfulness Questionnaire - 15 (FFMQ-15; Baer et al., 2006).
Subjective cognitive function (PDQ-D) | Development from pre-treatment to post-treatment and development from pre-treatment through 3-month follow-up
  Perceived Deficits Questionnaire - Depression (PDQ-D; Fehnel et al., 2016)
Experience of therapy | Session by session development during the 6 weeks of active treatment and through 3-month follow-up
  Five questions concerning the participants' experience or expectations concerning the components have been developed by the project group due to a lack of such assessment in the field.
Working alliance (WAI-SR) | Session 3 and 5 only
  Working Alliance Inventory - Short Revised (WAI-SR; Munder et al., 2010).
Information overload (IO) | Session by session development during the 6 weeks of active treatment
  The Information Overload (IO) scale, consisting of 8 items. This is our own adaptation of the Cancer Information Overload scale (Jensen et al., 2014) to assess perceived information overload related to the received treatment. This is included in all session questionnaires.

OTHER OUTCOMES:
Clinical diagnosis (ADIS-5) | Baseline only
  The Anxiety and Related Disorders Interview Schedule for DSM-5 (ADIS-5; Brown & Barlow, 2014) will be used to confirm a diagnosis of an anxiety disorder or MDD and establish the number of episodes, onset age, and potential comorbid disorders. The interview will also be used to confirm that none of the above listed reasons for exclusion are present (e.g., bipolar disorder, current or past psychosis).
Objective cognitive function - processing speed (TMT-A) | Baseline only
  Trail Making Test part A (TMT-A; Reitan, 1958).
Objective cognitive function - processing speed (WAIS-IV coding) | Baseline only
  Wechsler Adult Intelligence Scale - Fourth Edition, Coding (WAIS-IV coding; Wechsler, 2008).
Objective cognitive function - attention and working memory (WAIS-IV Digit span) | Baseline only
  Wechsler Adult Intelligence Scale - Fourth Edition, Digit span (WAIS-IV Digit span; Wechsler, 2008).
Objective cognitive function - executive function (COWAT) | Baseline only
  Controlled Oral Word Association Test (COWAT; Harrison et al., 2000).
Objective cognitive function - executive function (TMT-B) | Baseline only
  Trail Making Test part B (TMT-B; Reitan, 1958).
Objective cognitive function - executive function (STROOP) | Baseline only
  The Stroop Color and Word Test (STROOP; Stroop, 1935).
Objective cognitive function - premorbid intellectual abilities (WAIS-IV Information) | Baseline only
  Wechsler Adult Intelligence Scale - Fourth Edition, Information (WAIS-IV Information; Wechsler, 2008) will be included to control for premorbid intellectual abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Nørskov, MSc, Principal Investigator — University of Aarhus
Locations (1):
- Department of Psychology and Behavioral Sciences, Aarhus, Denmark

DOCUMENTS (2):
  • Statistical Analysis Plan: Original (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT06429956/SAP_000.pdf
  • Statistical Analysis Plan: Addition (2025-11-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT06429956/SAP_001.pdf